CLINICAL TRIAL: NCT04050722
Title: Randomized, Examiner Blind, Clinical Study Investigating the Efficacy of a Stannous Fluoride Dentifrice in Improving Gingival Health After 3 Weeks Use
Brief Title: A Clinical Study Investigating the Efficacy of a Stannous Fluoride Dentifrice in Improving Gingival Health After Twice Daily Use for 3 Weeks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 212537
Record Dates: First submitted 2019-08-07; First posted 2019-08-08 (Actual); Results first posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-10

CONDITIONS: Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single Blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Test Product (Experimental): Participants with no visible plaque will be instructed to apply full ribbon of the test product (containing 0.454 percent [%] of stannous fluoride] on head of toothbrush provided and brush their teeth for 1 timed minute twice a day (morning and evening), for 3 weeks.
  Interventions: Drug: Sensodyne Repair and Protect
- Negative Control Dentifrice (Other): Participants with no visible plaque will be instructed to apply full ribbon of the negative control dentifrice (containing sodium fluoride) on head of toothbrush provided and brush their teeth for 1 timed minute twice a day (morning and evening), for 3 weeks.
  Interventions: Drug: Colgate Cavity Protection

INTERVENTIONS:
Drug: Sensodyne Repair and Protect — Participants will brush their teeth with Sensodyne Repair and Protect (containing 0.454% stannous fluoride) for 1 timed minute twice a day (morning and evening), for 3 weeks.
  Arms: Test Product
Drug: Colgate Cavity Protection — Participants will brush their teeth with Colgate Cavity Protection repair and protect (containing sodium fluoride) for 1 timed minute twice a day (morning and evening), for 3 weeks.
  Arms: Negative Control Dentifrice

SUMMARY:
The aim of this study is to investigate the impact of a stannous fluoride containing toothpaste in reducing gingivitis when used twice daily for a maximum for 3 weeks, when compared to a standard sodium fluoride toothpaste (negative control).

DETAILED DESCRIPTION:
This will be a single center, controlled, single blind (examiner blind), randomized, two-treatment arm, parallel design, clinical study in participants (aged 18-65 years), with good general health (non-smokers) and generalized mild-moderate plaque-induced gingivitis and greater than equal to (>=) 20 natural teeth. The study consists of 4 study visits. At Visit 1, Screening, after signing informed consent, participants will be assessed for eligibility based on the inclusion/exclusion criteria and will undergo oral soft tissue (OST) and oral hard tissue (OHT) assessments. Participants will return between 1 and 28 days following the screening visit for the Visit 2, baseline where they will undergo, a full OST examination followed by assessments of gingival inflammation (MGI), gingival bleeding (BI) and supra-gingival plaque (TPI). Eligible participants will be stratified based on gender and baseline mean whole mouth MGI score (low: less than equal to (<=) 2.00/High greater than (>) 2.00), to ensure a balance of gingivitis across both treatment groups and then randomized to study product. All randomized participants will receive full mouth dental prophylaxis (followed by flossing) to remove sub and supra-gingival calculus, stain, plaque and debris from the teeth. All participants will enter the treatment period with no visible plaque (TPI=0). After all clinical assessments, participants will be instructed to brush for 1 timed minute at site with their assigned study product, after which they will be instructed to continue using this twice daily (morning and evening) for 2 weeks. After 2 weeks the participants will return to site for their Week 2 (Visit 3) assessments. They will then continue using their test dentifrice for a further week and will continue to record all brushing events in the diary provided, after which they will return for their Week 3 (Visit 4) assessments. All assessments will be carried out on the facial and lingual/palatal surfaces of each incisor, canine, pre-molar and molar, excluding third molars. After the Week 3 visit, study closeout procedures will take place and the participant may undergo an additional prophylaxis if it is deemed necessary by the examiner. Adverse events and incidents will be recorded from informed consent and at the end of each study visit.

ELIGIBILITY:
Inclusion Criteria:

An individual must meet all the following inclusion criteria to be eligible for enrollment into the study:

* Participant provision of a signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* A participant who is willing and able to comply with scheduled visits, treatment plan and other study procedures.
* A participant in good general and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant or relevant abnormalities in medical history or upon oral examination, or condition, that would impact the participant's safety, wellbeing or the outcome of the study, if they were to participate in the study, or affect the individual's ability to understand and follow study procedures and requirements.
* A participant at screening (Visit 1) with: a)at least 20 natural permanent teeth excluding 3rd molars; b)at least 40 evaluable surfaces (an evaluable surface is defined as having 2/3rds of the natural tooth surface gradable for the selected clinical indices. The following should not be included in the evaluable surface count- third molars; fully crowned/extensively restored, grossly carious, orthodontically banded/bonded or abutment teeth; surfaces with calculus deposits which, in the opinion of the clinical examiner, would interfere with the baseline assessments of the selected clinical indices); or c) participants with generalized mild-moderate plaque-induced gingivitis, in the opinion of the clinical examiner, as confirmed by visual examinations.
* A participant at baseline (prior to dental prophylaxis, (Visit 2) with: a)ongoing hard tissue eligibility and, in the opinion of the clinical examiner, at least 40 evaluable surfaces; b) mean whole mouth Modified Gingival Index (MGI) greater than equal to (>=) 1.75 to less than equal to (<=) 2.30; c) mean whole mouth supra-gingival Turesky Plaque Index (TPI) score ≥ 1.5; d) ≥ 20 bleeding sites.

Exclusion Criteria:

An individual who meets any of the following exclusion criteria will not be eligible for enrollment into the study:

* A participant who is an employee of the investigational site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the investigational site otherwise supervised by the investigator; or, a GlaxoSmithKline employee directly involved in the conduct of the study or a member of their immediate family.
* A participant who has participated in other studies (including non-medicinal studies) involving investigational product(s) within 30 days prior to study entry and/or during study participation.
* A participant with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the participant inappropriate for entry into this study.
* A participant with, in the opinion of the investigator or medically qualified designee, any clinically significant/relevant abnormalities in medical history or oral examination, or any other condition, that would affect the individual's ability to understand and follow study procedures and requirements.
* A participant with any medical condition which, in the opinion of the investigator or medically qualified designee, is causing xerostomia.
* A participant with any medical condition which in the opinion of the investigator or medically qualified designee, could directly influence gingival bleeding.
* A participant who is pregnant or intending to become pregnant over the duration of the study (self-reported).
* A participant who is breastfeeding.
* A participant with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* A participant with recent history (within the last year) of alcohol or other substance abuse.
* A participant who is a current smoker or an ex- smoker who stopped within 6 months of Screening.
* A participant who currently uses smokeless forms of tobacco (e.g. chewing tobacco, gutkha, pan containing tobacco, nicotine-based e-cigarettes).
* A participant with a severe oral condition (e.g. acute necrotizing ulcerative gingivitis or oral or peri-oral ulceration including herpetic lesions) that would, in the opinion of the investigator, compromise study outcomes or the oral health of the participant/ examiner if they were to participate in the study.
* A participant who has presence of a tongue or lip piercing, or any other oral feature that could interfere with the usage of a toothbrush
* A participant who, in the opinion of the investigator or medically qualified designee, should not participate in the study.
* A participant unwilling or unable to comply with the following Lifestyle Considerations (Dental Product/Treatment and Oral Hygiene Restrictions): a) From Screening (Visit 1) to the participants' last study visit- i) a participant should not carry out any interproximal dental cleaning. Use of dental floss, toothpicks, waterpicks or inter-dental brushes is prohibited (except for the removal of impacted food with non-antimicrobial products only), ii)participants should not chew gum or consume any confectionery containing xylitol (e.g. sugar-free mints), iii)participants should delay any non-emergency dental treatment until after study completion (including dental prophylaxis); b) From Baseline (Visit 2) to the participants last study visit- participants should not use any other oral care products (e.g. dentifrices, toothbrushes, mouth rinse) than those provided during the study; c) Before clinical efficacy assessment visits: Baseline (Visit 2), Week 2 (Visit 3) and Week 3 (Visit 4)- i) participant's should refrain from oral hygiene procedures for 12 hours (+6 hours, -2 hours) before their visit and attend the study site with overnight plaque growth.
* A participant that has used an anti-bacterial mouthwash (e.g. chlorhexidine) or use of any oral care product that in the view of the investigator could interfere with plaque formation or measures of gingivitis, within 14 days of the Baseline visit.
* Periodontal Exclusions: a) participant with signs of active periodontitis; b) participant with gingivitis which, in the opinion of the investigator, is not expected to respond to treatment with an over-the-counter dentifrice; c) A participant who is receiving or has received treatment for periodontal disease (including surgery) within 12 months of Screening.
* Dental Exclusions: a) participant with active caries that could, in the opinion of the investigator, compromise study outcomes or the oral health of the participant if they were to participate in the study; b )participant with dentures (partial or full); c) participant with an orthodontic appliance (bands, appliances or fixed/ removable retainers); d) A participant who has received orthodontic therapy within 12 months of screening; e) participant with numerous restorations in a poor state of repair; f) participant with any dental condition (e.g. overcrowding) that could, in the opinion of the investigator, compromise study outcomes or the oral health of the participant if they were to participate in the study; g) participant who has had dental prophylaxis within 12 weeks of Screening, h) participant who has had teeth bleaching within 12 weeks of Screening; i) A participant with high levels of extrinsic stain or calculus deposits that might interfere with plaque assessments. - Medication Exclusions: a )at screening (Visit 1)- i)participant who requires antibiotics prior to dental prophylaxis or other dental procedures, ii) participant who is currently taking antibiotics, iii) participant who is currently taking an anti-inflammatory medication which, in the opinion of the Investigator, could affect gingival condition (e.g. ibuprofen), iv) participant who is currently taking anti-coagulant medication which, in the opinion of the Investigator, could affect gingival condition (e.g. warfarin), v) participant who is currently taking a systemic medication or traditional/herbal remedy which, in the opinion of the Investigator, could affect gingival condition (e.g. immunosuppressants such as cyclosporine, phenytoin, calcium channel blockers, aspirin therapy); b) at baseline (Visit 2)- i) participant who has taken antibiotics in the 14 days prior to baseline, ii) participant who has taken an anti-inflammatory medication in the 14 days prior to baseline which, in the opinion of the Investigator, could affect gingival condition (e.g. ibuprofen), iii)participant who has taken anti-coagulant medication in the 14 days prior to Baseline which, in the opinion of the Investigator, could affect gingival condition (e.g. warfarin), iv)participant who has taken a systemic medication or traditional/herbal remedy in the 14 days prior to Baseline which, in the opinion of the Investigator, could affect gingival condition (e.g. immunosuppressants such as cyclosporine, phenytoin, calcium channel blockers, aspirin therapy), v) participant who has used an antibacterial dentifrice or mouth rinse in the period between Screening and Baseline.
* Any participant who has previously been enrolled in this study.
* Participants who, in the judgement of the investigator, or medically qualified designee should not participate on the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Acherkouk A, Patel N, Butler A, Amini P. A randomised clinical study investigating efficacy of a stannous fluoride toothpaste in improving gingival health after 3 weeks' use. BMC Oral Health. 2021 Sep 12;21(1):441. doi: 10.1186/s12903-021-01727-5. PMID 34511098

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one center in United States.
Pre-assignment Details: A total of 154 participants were screened, of whom 130 were randomized for treatment, 17 were screen failures, 3 withdrew consent prior to randomization, and 4 were not randomized as sufficient participants were already enrolled in the study.
Groups:
- Sensodyne Repair and Protect (Test Dentifrice): Participants randomized to this group brushed their teeth with Sensodyne Repair and Protect containing 0.454 percent (%) stannous fluoride (SnF2) (1100 parts per million [ppm] fluoride) for 1 timed minute twice a day (morning and evening) in their usual manner for 3 weeks. Participants recorded each brushing event in their dairy along with, any changes to these brushing procedures along with reasons for changes (e.g., missed brushings, extra brushings) and the actual time of the last brushing before attending site, on the day before the next visit.
- Colgate Cavity Protection (Negative Control Dentifrice): Participants randomized to this group brushed their teeth with Colgate Cavity Protection containing 1100 ppm fluoride as sodium monofluorophosphate (SMFP) for 1 timed minute twice a day (morning and evening) in their usual manner for 3 weeks. Participants recorded each brushing event in their dairy along with, any changes to these brushing procedures along with reasons for changes (e.g., missed brushings, extra brushings) and the actual time of the last brushing before attending site, on the day before the next visit.
Period: Overall Study
Arm/Group | Sensodyne Repair and Protect (Test Dentifrice) | Colgate Cavity Protection (Negative Control Dentifrice)
Started | 65 | 65
Completed | 64 | 65
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received at least one dose of the study product.
Groups:
- Sensodyne Repair and Protect (Test Dentifrice): Participants randomized to this group brushed their teeth with Sensodyne Repair and Protect containing 0.454 % SnF2 (1100 ppm fluoride) for 1 timed minute twice a day (morning and evening) in their usual manner for 3 weeks. Participants recorded each brushing event in their dairy along with, any changes to these brushing procedures along with reasons for changes (e.g., missed brushings, extra brushings) and the actual time of the last brushing before attending site, on the day before the next visit.
- Colgate Cavity Protection (Negative Control Dentifrice): Participants randomized to this group brushed their teeth with Colgate Cavity Protection containing 1100 ppm fluoride as SMFP for 1 timed minute twice a day (morning and evening) in their usual manner for 3 weeks. Participants recorded each brushing event in their dairy along with, any changes to these brushing procedures along with reasons for changes (e.g., missed brushings, extra brushings) and the actual time of the last brushing before attending site, on the day before the next visit.
- Total: Total of all reporting groups
Arm/Group | Sensodyne Repair and Protect (Test Dentifrice) | Colgate Cavity Protection (Negative Control Dentifrice) | Total
Number analyzed (Participants) | 65 | 65 | 130
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.3 (11.50) | 39.6 (12.48) | 39.4 (11.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 40 | 79
  Male | 26 | 25 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 15 | 34
  Not Hispanic or Latino | 46 | 50 | 96
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 6 | 10
  Native Hawaiian or Other Pacific Islander | 1 | 3 | 4
  Black or African American | 15 | 19 | 34
  White | 39 | 32 | 71
  More than one race | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Whole Mouth Mean Bleeding Index (BI) at Week 3
Description: BI method used to assess gingival bleeding as measure of gingival health for facial and lingual/palatal gingival surfaces of all evaluable teeth, six sites per tooth (mesiobuccal, buccal, distobuccal, mesiolingual/palatal, lingual/palatal, and distolingual/palatal). Examiner inserted a round-end probe approximately(app.) 1millimeter(mm) into gingival sulcus (at app 60 degrees) and moved around tooth, from distal interproximal area to mesial interproximal area, gently stretching gingival epithelium. Gingival bleeding was assessed 30 seconds after probing. Assessments performed 1 quadrant at a time; BI scores recorded as per given scoring criteria: 0=absence of bleeding on probing,1=bleeding observed within 30 seconds of probing,2=bleeding observed immediately on probing. Lower scores indicate better results. Mean whole mouth BI score for each participant was derived from total BI score divided by number of tooth sites scored. Overall mean calculated for all participants was reported.
Time Frame: Week 3
Population: Modified intent-to-treat (m-ITT) population was defined as all participants who were randomized, received at least one dose of the study treatments and provided at least one post-baseline assessment of efficacy. Here, number of participants analyzed indicates participants with available data for this outcome measure at specified time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sensodyne Repair and Protect (Test Dentifrice) | Colgate Cavity Protection (Negative Control Dentifrice)
Number analyzed (Participants) | 64 | 64
score on a scale | 0.14 (0.071) | 0.20 (0.066)
Statistical Analysis 1: Comparison: Sensodyne Repair and Protect (Test Dentifrice) vs Colgate Cavity Protection (Negative Control Dentifrice); Test type: Superiority; p < 0.0001, ANCOVA — Analysis was performed using ANCOVA model with study product group, gender, and baseline MGI stratification (low/high) as factors and the baseline value as covariate; Adjusted Mean Difference = -0.06, 95% CI 2-sided [-0.08 to -0.04], Standard Error of Mean 0.010

2. Secondary Outcome: Whole Mouth Mean Bleeding Index (BI) at Week 2
Description: BI method used to assess gingival bleeding as a measure of gingival health for facial and lingual/palatal gingival surfaces of all evaluable teeth, six sites per tooth (mesiobuccal, buccal, distobuccal, mesiolingual/palatal, lingual/palatal, and distolingual/palatal). Examiner inserted a round-end probe app. 1 mm into gingival sulcus (at app. 60 degrees) and moved around tooth, from distal interproximal area to mesial interproximal area, gently stretching gingival epithelium. Gingival bleeding was assessed 30 seconds after probing. Assessments were performed 1 quadrant at a time; BI scores were recorded as per given scoring criteria: 0=absence of bleeding on probing,1=bleeding observed within 30 seconds of probing,2=bleeding observed immediately on probing. Lower scores indicate better results. Mean whole mouth BI score for each participant was derived from total BI score divided by number of tooth sites scored. Overall mean calculated for all participants was reported.
Time Frame: Week 2
Population: m-ITT population was defined as all participants who were randomized, received at least one dose of the study treatments and provided at least one post-baseline assessment of efficacy.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sensodyne Repair and Protect (Test Dentifrice) | Colgate Cavity Protection (Negative Control Dentifrice)
Number analyzed (Participants) | 64 | 65
score on a scale | 0.15 (0.072) | 0.22 (0.073)

3. Secondary Outcome: Mean Number of Bleeding Sites (NBS) at Week 2 and Week 3
Description: Number of bleeding sites were derived from the bleeding index (BI). BI method used to assess gingival bleeding as a measure of gingival health for facial and lingual/palatal gingival surfaces of all evaluable teeth, six sites per tooth (mesiobuccal, buccal, distobuccal, mesiolingual/palatal, lingual/palatal, and distolingual/palatal). Examiner inserted a round-end probe app. 1 mm into gingival sulcus (at app. 60 degrees) and moved around tooth, from distal interproximal area to mesial interproximal area, gently stretching gingival epithelium. Gingival bleeding was assessed 30 seconds after probing. Assessments were performed 1 quadrant at a time; BI scores were recorded as per given scoring criteria: 0=absence of bleeding on probing,1=bleeding observed within 30 seconds of probing,2=bleeding observed immediately on probing. Lower scores indicate better results. A bleeding site was a site scored as 1 or 2. Mean of all bleeding sites was calculated and reported.
Time Frame: Week 2 and Week 3
Population: m-ITT population was defined as all participants who were randomized, received at least one dose of the study treatments and provided at least one post-baseline assessment of efficacy. Here, number analyzed indicates participants with available data at specified time point.
Measure: Mean (Standard Deviation); unit: number of bleeding sites
Arm/Group | Sensodyne Repair and Protect (Test Dentifrice) | Colgate Cavity Protection (Negative Control Dentifrice)
Number analyzed (Participants) | 64 | 65
number of bleeding sites
  At Week 2 | 21.0 (10.14) | 31.7 (10.93)
  At Week 3: number analyzed (Participants) | 64 | 64
  At Week 3 | 19.7 (10.17) | 28.0 (9.60)

4. Secondary Outcome: Mean Modified Gingival Index (MGI) at Week 2 and Week 3
Description: MGI used to assess for visual symptoms of gingivitis (redness, texture, edema) for all evaluable teeth, four sites per tooth (facial surface - papilla and margin; lingual/palatal surface - papilla and margin). MGI scores were recorded as per given scoring criteria: 0- Absence of inflammation, 1- Mild inflammation: slight change in color, little change in texture of any portion of marginal or papillary gingival unit, 2- Mild inflammation: criteria as [1] but involving entire marginal or papillary gingival unit, 3- Moderate inflammation: glazing, redness, edema, and/or hypertrophy of marginal or papillary gingival unit, 4- Severe inflammation: marked redness, edema and/or hypertrophy of marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration. Lower scores indicate better results. Mean whole mouth MGI score for each participant was derived from total MGI score divided by number of tooth sites scored. Overall mean calculated for all participants was reported.
Time Frame: Week 2 and Week 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sensodyne Repair and Protect (Test Dentifrice) | Colgate Cavity Protection (Negative Control Dentifrice)
Number analyzed (Participants) | 64 | 65
score on a scale
  At Week 2 | 2.08 (0.142) | 2.18 (0.113)
  At Week 3: number analyzed (Participants) | 64 | 64
  At Week 3 | 2.05 (0.152) | 2.15 (0.124)

5. Secondary Outcome: Mean Overall Turesky Modification of the Quigley & Hein Plaque Index (TPI) Score at Week 2 and Week 3
Description: TPI assessed supra-gingival plaques on facial and lingual surfaces of all evaluable teeth. Each tooth divided into 3 areas;3 scores recorded facially (mesiofacial,facial,distofacial) and 3 scores lingually (mesiolingual,lingual,distolingual) generating a total of 6 scores per tooth. Plaque was identified using disclosing solution followed by rinsing with tap water(10 milliliters for 10 seconds) and scored as per given scoring criteria:0-no plaque,1-separate flecks of plaque at cervical margin,2-thin continuous band of plaque (up to 1mm) at cervical margin,3-band of plaque wider than 1mm but covering less than(<)1/3 of tooth surface,4-plaque covering more than or equal to (>=)1/3 but <2/3 of tooth surface,5-plaque covering >=2/3 of tooth surface. Lower scores indicate better results. Mean Overall TPI score for each participant was derived from total TPI score over all tooth sites divided by number of tooth sites scored. Overall mean calculated for all participants was reported.
Time Frame: Week 2 and Week 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sensodyne Repair and Protect (Test Dentifrice) | Colgate Cavity Protection (Negative Control Dentifrice)
Number analyzed (Participants) | 64 | 65
score on a scale
  At Week 2 | 2.35 (0.333) | 2.81 (0.307)
  At Week 3: number analyzed (Participants) | 64 | 64
  At Week 3 | 2.33 (0.420) | 2.76 (0.303)

6. Secondary Outcome: Mean Interproximal Turesky Modification of the Quigley & Hein Plaque Index (TPI) at Week 2 and Week 3
Description: TPI assessed supra-gingival plaques on facial and lingual surfaces of all evaluable teeth. Each tooth was divided into 3 areas; 3 scores were recorded facially (mesiofacial,facial,distofacial) and 3 scores lingually (mesiolingual,lingual,distolingual) generating a total of 6 scores per tooth. Plaque was identified using disclosing solution followed by rinsing with tap water(10 milliliters for 10 seconds) and scored as per given scoring criteria: 0-no plaque,1-separate flecks of plaque at cervical margin,2-thin continuous band of plaque(up to 1 mm)at cervical margin,3-band of plaque wider than 1mm but covering <1/3 of tooth surface,4-plaque covering >=1/3 but <2/3 of tooth surface,5-plaque covering >=2/3 of tooth surface. Lower scores indicate better results. Mean Interproximal TPI score for each participant was derived from total TPI score over all interproximal tooth sites divided by number of interproximal tooth sites scored. Mean calculated for all participants was reported.
Time Frame: Week 2 and Week 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sensodyne Repair and Protect (Test Dentifrice) | Colgate Cavity Protection (Negative Control Dentifrice)
Number analyzed (Participants) | 64 | 65
score on a scale
  At Week 2 | 2.48 (0.338) | 2.90 (0.279)
  At Week 3: number analyzed (Participants) | 64 | 64
  At Week 3 | 2.47 (0.421) | 2.88 (0.273)

ADVERSE EVENTS:
Time Frame: Up to 28 days
Description: Safety population included all randomized participants who received at least one dose of the study product.All adverse events (AEs) were summarized by system organ class and preferred term. All treatment emergent AEs and serious adverse events (SAEs) were collected and reported. A participant with multiple occurrences of AEs counted once in AE category. A participant with multiple AEs within a primary system organ class was counted once in system organ class.
Arm/Group | Sensodyne Repair and Protect (Test Dentifrice) | Colgate Cavity Protection (Negative Control Dentifrice)
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/65
Other Adverse Events (participants affected / at risk) | 4/65 | 3/65
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sensodyne Repair and Protect (Test Dentifrice) (N=65) | Colgate Cavity Protection (Negative Control Dentifrice) (N=65)
Gingival injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Traumatic ulcer (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gingival ulceration (Gastrointestinal disorders) | 0 (0) | 1 (3)
Angular cheilitis (Infections and infestations) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-06-22): https://cdn.clinicaltrials.gov/large-docs/22/NCT04050722/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-04): https://cdn.clinicaltrials.gov/large-docs/22/NCT04050722/SAP_001.pdf